CLINICAL TRIAL: NCT04686734
Title: Long-term Effects of COVID-19 in Adolescents
Acronym: LoTECA
Status: Completed | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Vegard Wyller, Professor, University Hospital, Akershus
Other Study IDs: LoTECA
Record Dates: First submitted 2020-12-27; First posted 2020-12-29 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SARS-CoV-2 positive
  Interventions: Other: No active intervention (observational only)
- SARS-CoV-2 negative
  Interventions: Other: No active intervention (observational only)

INTERVENTIONS:
Other: No active intervention (observational only) — No active intervention (observational only)

SUMMARY:
The overarching objective for this prospective cohort study of COVID-19 in adolescents is to study the long-term effects, with particular emphasis on post-infectious chronic fatigue. A total of 500 individuals with a SARS-CoV-2 positive test will be enrolled in the acute phase of COVID-19 and followed for 6 months. A total of 100 individuals with SARS-CoV-2 negative test will be included during the same time period as a control group. Investigations include autonomic, pulmonary and cognitive assessement; a questionnaire charting symptoms, emotionality, personality, loneliness, life events and demographics; and extensive biobanking including genetic markers, viable PBMC, urine, feces and hair. A subgroup of 40 SARS-CoV-2 positive and 20 SARS-CoV-2 negative individuals will also undergo detailed cardiological examination by echocardiography. Primary endpoints are fatigue at 6 months as assessed by the Chalder Fatigue Scale and post-COVID-19 syndrome cases at 6 months according to the WHO definition

ELIGIBILITY:
Inclusion Criteria:

* Positive SARS-CoV-2 test/negative SARS-CoV-2 test
* Age 12 - 25 years
* Living in the counties of Oslo or Viken, Norway
* < 28 days since onset of first symptom

Exclusion Criteria:

* Hospitalised due to COVID-19
* Pregnancy
* Lack of consent

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents living in the counties of Oslo and Viken, Norway
Sampling Method: Non-Probability Sample
Enrollment: 516 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Fatigue | 6 months follow-up
  Total sum score on the Chalder Fatigue Scale (range 0 - 33, lower scores means less fatigue, ie. better outcome)
Post-COVID-19 syndrome caseness | 6 months follow-up
  Post-COVID-19 syndrome casesness according to the WHO definition (issued Sept. 2021; hence, this endpoint was added during the course of the study, but prior to database lock.)

CONTACTS AND LOCATIONS:
Overall Officials: Vegard B Wyller, PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Vegard Bratholm Wyller, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lund Berven L, Selvakumar J, Havdal L, Stiansen-Sonerud T, Einvik G, Leegaard TM, Tjade T, Michelsen AE, Mollnes TE, Wyller VBB. Inflammatory Markers, Pulmonary Function, and Clinical Symptoms in Acute COVID-19 Among Non-Hospitalized Adolescents and Young Adults. Front Immunol. 2022 Feb 9;13:837288. doi: 10.3389/fimmu.2022.837288. eCollection 2022. PMID 35222429
- See also: Information for patients and other public stakeholders — https://www.ahus.no/kliniske-studier/langtidseffekter-etter-koronavirusinfeksjon-covid-19-hos-ungdommer

DOCUMENTS (2):
  • Study Protocol (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/34/NCT04686734/Prot_003.pdf
  • Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/34/NCT04686734/SAP_004.pdf